CLINICAL TRIAL: NCT03883217
Title: Optimizing Vibrational Therapy to Improve Gait and Balance in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HM20015593
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Gait; Balance
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Vibration first then no vibration (Experimental): A session with PDVibe2 vibration turned on first, followed by (after a 2 week washout period) a session with PDVibe2 vibration turned off.
  Interventions: Device: PDVibe2
- No vibration first then vibration (Experimental): A session with PDVibe2 vibration turned off first, followed by (after a 2 week washout period) a session with PDVibe2 vibration turned on.
  Interventions: Device: PDVibe2

INTERVENTIONS:
Device: PDVibe2 — The PDVibe2 is owned by Resonate Forward, LLC and will be loaned to Virginia Commonwealth University (VCU) for this project. The device is non-invasive, lightweight, untethered, contains a rechargeable battery, and is worn on both feet and ankles. PDVibe2 delivers vibration when activated by an easy to access switch on the device or by remote. The internal circuitry has been miniaturized, is encased in a small box, and is attached to the ankle using a soft flexible band.
  Other Names: VibeForward

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and the effect of vibration (delivered by an experimental device called PDVibe2) on freezing of gait (FOG) in persons with Parkinson's disease (PD). The PDVibe2 was developed by Resonate Forward, LLC (RF). This PDVibe2 was designed to administer vibration therapy to the wearer to improve gait and balance in persons with PD while wearing the device.

DETAILED DESCRIPTION:
Enrolled patients with Parkinson's disease, Hoehn and Yahr Stage 2, will be randomized to receive either vibration or no vibration and then will be crossed over to receive the opposite intervention. The study will consist of two treatment periods of two days followed by a washout period of 2 weeks. Each treatment period will consist of four treatments within 2 days, no more than 2 sessions in one day.

Patients will participate in an additional day for screening and another for follow-up (6 days total). All visits will occur at the Virginia Commonwealth University Parkinson's Movement and Disorders Center in Richmond, VA. Participants will be asked to walk for a brief period of time while wearing the PDVibe2. The PDVibe2 will provide vibration therapy and study staff will measure the number of "freezes" before, during and after therapy. Participants will be asked to provide feedback on the device, the therapy session, and how they are feeling.

ELIGIBILITY:
Inclusion criteria:

* age 21 years or older
* PD diagnosed by a movement disorder specialist for 3 months or longer prior to recruitment
* PD medication regimen is stable over the last 3 months with no changes
* Hoehn & Yahr stage 2 (N = 13)
* able to walk independently or with a simple assistive device (e.g., cane, walker)
* observed by the research team to have PD related gait disturbance such as FOG, shortened or irregular stride lengths, irregular step cadence, slowed speed while on their regular treatment regimen.

Exclusion Criteria:

* diagnosed with a known Parkinson plus syndrome
* were previously exposed to vibration treatment for gait and balance
* presence of dementia (Montreal Cognitive Assessment < 21)
* additional disorders (not related to PD)impairing gait, stance, balance or coordination (e.g. stroke, leg amputations, or multiple sclerosis)
* history of implantable cardiac device or any other implanted electronic device except a deep brain stimulator (DBS)
* use of braces/orthotics that assist with walking
* are currently in physical therapy (PT) treatment for balance or gait
* peripheral neuropathy by exam
* any condition that, in the opinion of the PIs, would compromise participant safety, data integrity, or data interpretation.
* Children under the age of 18
* Prisoners
* Women who are pregnant or may become pregnant during the course of this study since the safety of this device for an unborn child is unknown.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Profile (FAP) Score | Throughout study completion, from 9 to 34 days.
  The FAP score is the gold standard for spatiotemporal gait parameter analysis. For this study, it will be calculated by participants walking on the Zeno walkway, which will measure the patient's physical measurements, step length, step time and degree of symmetry.Step length, step time, degree of symmetry, dynamic base of support and the use of ambulatory aids are factored into the score. The Zeno instrumented walkway (PKMAS) is a 20-foot computerized instrumented walkway containing sensor pads.

SECONDARY OUTCOMES:
Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) Part III | Throughout study completion, between 9 to 34 days.
  The "Movement Disorder Society Unified Parkinson Disease Rating Scale" (MDS-UPDRS), parts II-IV will be used to assess the total burden of motor Parkinson Disease (PD) symptoms and impact on activities of daily living. All parts use scale of 0 (no problem) - 4 (severe problems) lower scores are better. Part II: 13 items about Activities of Daily Living, score range 0-52. Part III: 18 items PD motor signs, score range is 0-72, Part IV: 6 items, assesses dyskinesia (excessive motion) and motor fluctuations (medication is working or not), range is 0-24. Parts II-IV total scores will be summed and used to describe the participants, total score range 0-148. Part III, only, will be repeated during vibration and post vibration data collection times and will take 5 minutes to complete. This outcome measure will be used to report a change in PD motor symptoms from baseline, to vibration on, and at follow up two after treatment is completed.
Timed Up and Go (TUG) Test | Throughout study completion, between 9 to 34 days.
  This test is a one item performance test. The participant starts by sitting in a chair, then stand up, walk 3 meters, turn around, walk back, and sit down. Participants are timed in seconds. TUG is used to identify/screen elderly individuals who are prone to falls. Lower numbers are better.
Berg Balance Scale (BBS) | Throughout study completion, between 9 to 34 days.
  The BBS assesses balance via performing 14 functional activities. Each item is scored along a 5-point scale, ranging from 0 to 4. Zero indicates the lowest level of function and 4 the highest level of function. The total score is a summation of all items and ranges from 0 to 56. Higher scores indicate less risk of falls. A cutoff score of 45 has been traditionally identified as a useful cutoff to predict falls in those who scored below the cutoff score.
Freezing of Gait Questionnaire (FOG-Q) | Throughout study completion, between 9 to 34 days
  The FOG-Q is a six-item questionnaire that uses a 5-point scale that ranges from 0 = absence of symptoms to 4 = most severe stage. The total score ranges from 0 to 24; higher scores correspond to more severe FOG.
Fall Efficacy Scale - International | Throughout study completion, between 9 to 34 days.
  This survey includes 16 items assessing fear of falling in different scenarios, in a community dwelling older population. Individuals are instructed to rate each activity on a four-point Likert scale, depending on how they concerned that they may fall when performing certain activities. Items are scored from 1 = Not at all concerned to 4 = very concerned. The total score ranges from 16 - 64. The higher the score the greater the fear of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Pretzer-Aboff, PhD, RN, Principal Investigator — Virginia Commonwealth University; Leslie Cloud, MD, Principal Investigator — Virginia Commonwealth University Health System
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No